CLINICAL TRIAL: NCT06348407
Title: The Efficacy and Safety of Omalizumab in the Treatment of Moderate to Severe Allergic Asthma:A Retrospective Single-center Clinical Trial
Brief Title: A Clinical Study of Omalizumab in the Treatment of Allergic Asthma(ESSENCE)
Acronym: ESSENCE
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-BA-001
Record Dates: First submitted 2024-03-21; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Moderate to Severe Allergic Asthma
Keywords: asthma; omalizumab; allergy; IgE
MeSH Terms: conditions — Asthma; Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Responder group: The improvement in ACT score ≥ 3,or pre-treatment ACT score < 20 and a post-treatment ACT score ≥ 20；The GETE score was excellent or good.
  Interventions: Drug: IgE monoclonal antibody
- No-Responder group: The improvement in ACT score < 3;The GETE score was moderate,poor and worse.
  Interventions: Drug: IgE monoclonal antibody
- Good adherence: The proportion of patients whose missed doses of omalizumab fewer than 10% of all doses over the1 year, we think these patients were good adherence.
  Interventions: Drug: IgE monoclonal antibody
- Poor adherence: the proportion of patients who missed at least 10% of all doses over the 1year,we think these patients were poor adherence.
  Interventions: Drug: IgE monoclonal antibody

INTERVENTIONS:
Drug: IgE monoclonal antibody — omalizumab

SUMMARY:
Allergic asthma being the most widespread and easily identifiable phenotype, accounting for 60-80% of cases.Previous studies have reported that nearly 90% of patients with severe asthma were cases of allergic asthma, in which Immunoglobulin E (IgE) plays a critical role.Omalizumab was approved as an anti-IgE humanized monoclonal antibody for the treatment of patients with poorly controlled moderate-to-severe asthma, and was the first targeted drug used in the field of asthma treatment.The drug was launched in mainland China in August 2017.whereas,the clinical application experience, effects, and relevant data in the domestic population still lacking.The aim of this study was to observe the efficacy and safety of omalizumab, and to investigate whether baseline clinical characteristics and biomarkers can predicted response and adherence to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Moderate-to-severe asthma patients aged ≥ 14 years who met the criteria of the Asthma Group of the Chinese Thoracic Society (Guidelines for bronchial asthma prevention and management, 2020 edition)-moderate asthma was defined as those who could achieve complete control using grade 3 therapy, and severe asthma was defined as fully or incompletely controlled with grade 4 or 5 asthma medications.
* History of asthma exacerbations induced by allergen exposure , elevated total serum IgE and positive specific IgE test or positive skin prick test.
* Treatment with omalizumab.

Exclusion Criteria:

* Hypersensitivity to the active ingredient of omalizumab.
* Asthma exacerbation in the baseline.
* Combined with diseases that severely affect ventilation,such as bronchiectasis, lung cancer, allergic bronchopulmonary aspergillosis (ABPA), acute respiratory infections, chronic obstructive pulmonary disease (COPD),etc.
* Receiving other biologically targeted therapies (e.g., anti-interleukin (IL)-5 monoclonal antibody, anti-IL-4 monoclonal antibody, anti-IL-13 monoclonal antibody, anti-IL-5 receptor α (IL-5Rα) monoclonal antibody, etc.)

Ages: 14 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with moderate to severe allergic asthma who received omalizumab at the First Affiliated Hospital with Nanjing Medical University from 2018 to 2023.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in Asthma Control Test (ACT) | Baseline, up to16weeks，24weeks and 1year of treatment.
  The responder in ACT was required to meet any of the following conditions:(a) an improvement in ACT score ≥ 3 (MID); and (b) a pre-treatment ACT score < 20 (poor or poorly controlled asthma) and a post-treatment ACT score ≥ 20 (well controlled asthma).
Global Evaluation of Treatment Effectiveness (GETE) | Baseline, up to16weeks，24weeks and 1year of treatment.
  Global Evaluation of Treatment Effectiveness (GETE) score after omalizumab treatment. The responder in GETE is score of "excellent" or"good" after treatment.

SECONDARY OUTCOMES:
Forced Expiratory Volume in 1 second（FEV1) | Baseline, up to 16weeks，24weeks and 1year of treatment.
  Pre-bronchodilators FEV1 .
FEV1/predicted%. | Baseline, up to 16weeks，24weeks and 1year of treatment.
  Pre-bronchodilators FEV1/predicted%.
Forced Vital Capacity （FVC） | Baseline, up to16weeks，24weeks and 1year of treatment.
  Pre-bronchodilators FVC
FEV1/FVC. | Baseline, up to16weeks，24weeks and 1year of treatment.
  Pre-bronchodilators FEV1/FVC.
Number of Acute Exacerbations（AE） | up to16weeks，24weeks and 1year of treatment.
  Number of acute exacerbations 1 year before omalizumab treatment,and up to16weeks，24weeks and 1year of treatment.
Oral glucocorticoid dosage | up to16weeks，24weeks and 1year of treatment.
  Oral glucocorticoid dosage before and after omalizumab treatment
Good adherence | 1 year
  Adherence to omalizumab treatment in this study was assessed by examining the rates of missed doses,the proportion of patients who missed fewer than 10% of all doses over 1 years was good adherence.
Poor adherence | 1 year
  Adherence to omalizumab treatment in this study was assessed by examining the rates of missed doses,the proportion of patients who missed at least 10% of all doses over 1 year was poor adherence.
Adverse events | up to16weeks，24weeks and 1year of treatment.
  Incidence of adverse events = Number of subjects with adverse events/Total number of subjects in treatment×100%

CONTACTS AND LOCATIONS:
Locations (1):
- Linfu zhou, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Protect patient privacy